CLINICAL TRIAL: NCT03012776
Title: A Clinical Study to Assess the Safety and Effectiveness of the Premia Spine TOPS™ System
Brief Title: A Pivotal Study of the Premia Spine TOPS™ System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Premia Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-2830 - US IDE
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lumbar Spinal Stenosis; Degenerative Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TOPS System (Experimental): Investigational surgical treatment using TOPS System
  Interventions: Device: Total Posterior Spine System (TOPS)
- Transforaminal Lumbar Interbody Fusion (TLIF) (Active Comparator): Control surgical treatment using interbody fusion and placement of posterolateral instrumentation
  Interventions: Procedure: Transforaminal Lumbar Interbody Fusion (TLIF)

INTERVENTIONS:
Device: Total Posterior Spine System (TOPS) — Placement of TOPS System to provide posterior stabilization following decompression to treat lumbar spinal stenosis and spondylolisthesis
  Arms: TOPS System
Procedure: Transforaminal Lumbar Interbody Fusion (TLIF) — Fusion with placement of interbody cage and posterolateral instrumentation
  Arms: Transforaminal Lumbar Interbody Fusion (TLIF)

SUMMARY:
The purpose of this trial is to assess whether the Total Posterior Spine System (TOPS System) is more effective than transforaminal lumbar interbody fusion (TLIF) when used to stabilize a single lumbar level (L2 - L5) following surgical decompression in patients diagnosed with (1) at least moderate lumbar spinal stenosis, and (2) Grade 1 spondylolisthesis (or retrolisthesis), and (3) thickening of the ligamentum flavum or scarring of the facet joint capsule.

Success will be assessed by means of a composite endpoint that measures improvement in in patient reported outcomes and the absence of any major device related complications.

DETAILED DESCRIPTION:
Degenerative spine disease is a normal part of the aging process and can cause pain and significantly limit normal movement. The most commonly diagnosed condition is Lumbar Spinal Stenosis (LSS) which presents with pain, and often weakness or numbness in the buttocks and/or lower extremities that is worsened with standing and walking. For patients that do not respond to conservative treatment decompressive surgery is indicated. When LSS is accompanied by a diagnosis of degenerative spondylolisthesis, fusion of the affected segment is often added to prevent progression of the instability that may accompany the removal of bony elements as part of the decompression. While decompression and fusion have been shown to significantly improve patient outcomes, when compared to decompression alone, fusion has been associated with several comorbidities such as adjacent level degeneration and pseudoarthrosis.

The TOPS System was designed as an alternative to fusion and is a motion preserving posterior spine implant designed to provide dynamic stabilization to a single lumbar spine segment following decompression surgery.

Patients meeting all of the entry criteria will be randomized (2:1) to receive either the TOPS System or TLIF following decompression surgery. Patients will be followed for 5 years and the composite primary endpoint will be assessed at 2 years following index surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be between 35 and 80 years of age;
* Must demonstrate at a single level to be treated (L2/3, L3/4 or L4/5) all three of the following;

  1. Degenerative spondylolisthesis or retrolisthesis up to Grade I, as determined by the investigator based on flexion/extension X-rays,
  2. At least moderate lumbar spinal stenosis, defined as at least a 25% reduction in either the central canal, the lateral recess space, and/or the foramen when compared to an adjacent level, as determined by the investigator based on MRI,
  3. Thickening of the ligamentum flavum and/or scarring of the facet joint capsule as identified by the investigator based on MRI.
* Have had at least six (6) months of failed conservative treatment prior to surgery (e.g., physical therapy, use of anti-inflammatory medications at maximum recommended dosage; administration of epidural/facet injections and/or nerve block);
* Have an Oswestry Disability Index (ODI) score of at least 40/100 at baseline;
* Have leg pain with a VAS score of at least 40/100 for at least one leg at baseline ;
* Lower back pain with a VAS score of at least 10 points less than Worst Leg VAS score;
* Neurogenic claudication (as defined by worsening leg pain when walking or standing, which is reduced when sitting or bending forward);

Exclusion Criteria:

* Presence of free fragment disc herniation at the index level or either adjacent level;
* Less than 4mm of disc height at the index level;
* Spondylolisthesis greater than Grade I;
* Back or non-radicular leg pain of unknown etiology;
* Stenosis caused by an extruded spinal disc fragment (e.g., herniation) or where the etiology is considered to be congenital, iatrogenic, post-traumatic, or metabolic;
* Known allergy or sensitivity to PEEK, titanium, cobalt chrome, and/or polyurethane;
* Prior surgery at any lumbar vertebral level with instrumentation;
* Prior surgery at the index or adjacent lumbar vertebral level;
* Clinically compromised vertebral bodies at the affected level;
* Scoliosis greater than ten (10) degrees by major Cobb angle;
* BMI > 40;
* Osteoporosis;
* Paget's disease, gout, osteomalacia, osteogenesis imperfecta, thyroid and/or parathyroid gland disorder and/or other metabolic bone disease;
* Active infection - systemic or local;
* Active hepatitis;
* AIDS, HIV, Rheumatoid arthritis or other autoimmune disease;
* Tuberculosis - active or in the past 3 years;
* Active malignancy;
* Any medical condition requiring treatment with any drug known to potentially interfere with bone/soft tissue healing or receiving radiation therapy that is expected to continue for the duration of the study;
* Cauda equina syndrome or neurogenic bowel/bladder dysfunction;
* Vascular claudication due to severe arterial insufficiency of the legs;
* Sustained pathologic lumbar fractures of the vertebra or multiple lumbar fractures of the vertebra or hip;
* Significant peripheral neuropathy causing decreased sensation in a stocking-like or non-radicular and non-dermatomal distribution in the lower extremities;
* Insulin-dependent diabetes mellitus;
* Immunologically suppressed, receiving steroids > 1 month out of the past year;
* Current chemical/alcohol dependency;
* Current smoker or user of tobacco products;
* Pregnant or interested in becoming pregnant;
* Currently involved in active spinal litigation;
* Currently having a workman's compensation claim;
* Currently incarcerated;

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Improvement in Oswestry Disability Index (ODI) | 24 months
Maintenance or improvement in Neurological status as assessed by a standard neurological exam performed by Investigator | 24 months
No epidural steroid injection, facet joint injection, nerve block, or placement of spinal cord stimulator | 24 months
No subsequent surgical intervention | 24 months
Radiographic confirmation of fusion in control arm and non-fusion in the TOPS arm | 24 months
Absence of any major device related adverse event | 24 months

SECONDARY OUTCOMES:
Greater range-of-motion through flexion-extension | 24 months
Improvement (20 mm) in visual analogue scale (VAS) for back pain and worst leg | 24 months
Reduction in physical component score on SF-12 | 24 months

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Adventist Health Glendale, Glendale, California
  - Cedars Sinai, Los Angeles, California
  - University of California - Irvine Medical Center, Orange, California
  - Eisenhower Desert Orthopedic Center, Palm Desert, California
  - St. Mary's Medical Center, Spine Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Boulder Neurosurgical & Spine Associates, Boulder, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Hospital/Johns Hopkins, Washington D.C., District of Columbia
  - Florida Spine Institute, Clearwater, Florida
  - St. Vincent's Spine & Brain Institute, Jacksonville, Florida
  - Physicians Regional Medical Center, Naples, Florida
  - Kennedy White Orthopedic Center, Sarasota, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Goodman Campbell Brain & Spine, Carmel, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Bronson Neuroscience Center, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Lenox Hill Hospital, New York, New York
  - Carolina Neurosurgery & Spine Associates, P.A., Charlotte, North Carolina
  - Univ. of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Southern Oregon Orthopedics, Medford, Oregon
  - Orthopedic Institute of Pennsylvania, Harrisburg, Pennsylvania
  - UPENN Health Systems Department of Neurosurgery, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Orthopaedic Associates, Bellaire, Texas
  - Texas Back Institute, Plano, Texas
  - Baylor Scott & White, Temple, Texas
  - Neurosurgical Associates, P.C., Richmond, Virginia
  - Marshall University, Huntington, West Virginia
  - Wisconsin Bone and Joint S.C., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coric D, Nassr A, Kim PK, Welch WC, Robbins S, DeLuca S, Whiting D, Chahlavi A, Pirris SM, Groff MW, Chi JH, Huang JH, Kent R, Whitmore RG, Meyer SA, Arnold PM, Patel AI, Orr RD, Krishnaney A, Boltes P, Anekstein Y, Steinmetz MP. Prospective, randomized controlled multicenter study of posterior lumbar facet arthroplasty for the treatment of spondylolisthesis. J Neurosurg Spine. 2022 Sep 23;38(1):115-125. doi: 10.3171/2022.7.SPINE22536. Print 2023 Jan 1. PMID 36152329